CLINICAL TRIAL: NCT02279420
Title: A Supplemental Open Label Multicenter Sham Cross-over Clinical Trial Using an Endoscopic Suturing Device (g-Cath EZ™ Suture Anchor Delivery Catheter) For Primary Weight Loss Essential Study (IDE G130163) Crossover Study
Brief Title: ESSENTIAL Trial™ Sham Cross-over
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPR 50402
Record Dates: First submitted 2014-10-23; First posted 2014-10-31 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Essential Study Sham Cross-over (Other): Device: g-Cath EZ™ Suture Anchor Delivery Catheter This is a multicenter, un-blinded, open label, pivotal supplemental study to G130163 intended to evaluate the safety and efficacy of treating previous sham subjects in the Essential pivotal trial (IDE#G130163) with the active treatment (the placement of g-Cath EZ suture anchors along with diet and exercise). Compliant sham subjects (those who attended all primary IDE follow-up visits AND who continue to meet eligibility criteria as described in this protocol) will be offered this active treatment after their 12 month unblinding visit in the Essential pivotal trial.
  Interventions: Device: g-Cath EZ™ Suture Anchor Delivery Catheter

INTERVENTIONS:
Device: g-Cath EZ™ Suture Anchor Delivery Catheter — This is a multicenter, un-blinded, open label, pivotal supplemental study to G130163 intended to evaluate the safety and efficacy of treating previous sham subjects in the Essential pivotal trial (IDE#G130163) with the active treatment (the placement of g-Cath EZ suture anchors along with diet and exercise). Compliant sham subjects (those who attended all primary IDE follow-up visits AND who continue to meet eligibility criteria as described in this protocol) will be offered this active treatment after their 12 month unblinding visit in the Essential pivotal trial.

SUMMARY:
This is a multicenter, un-blinded, open label, pivotal supplemental study to G130163 intended to evaluate the safety and efficacy of treating previous sham subjects in the Essential pivotal trial (IDE#G130163) with the active treatment (the placement of g-Cath EZ suture anchors along with diet and exercise). Compliant sham subjects (those who attended all primary IDE follow-up visits AND who continue to meet eligibility criteria as described in this protocol) will be offered this active treatment after their 12 month unblinding visit in the Essential pivotal trial.

DETAILED DESCRIPTION:
This is a multicenter, un-blinded, open label, pivotal supplemental study to G130163 intended to evaluate the safety and efficacy of treating previous sham subjects in the Essential pivotal trial (IDE#G130163) with the active treatment (the placement of g-Cath EZ suture anchors along with diet and exercise). Compliant sham subjects (those who attended all primary IDE follow-up visits AND who continue to meet eligibility criteria as described in this protocol) will be offered this active treatment after their 12 month unblinding visit in the Essential pivotal trial.

This supplemental study will consist of up to an 8 week screening period after each subject's unblinding visit, an enrollment (active treatment) day, and a 12-month follow-up period. All sham subjects in the Essential Trial (total quantity of one hundred eleven (111) subjects) are planned for enrollment, but the total quantity of sham subjects provided the active treatment will depend on the number of subjects who are compliant. The active treatment will be provided by the original investigator for that subject at the same investigational center (one of the original 11) used in the Essential trial. Collection of data will be accomplished by utilizing independent nutritionists/clinical research nurses to administer the diet/exercise plan and collect weight loss efficacy assessments. Efficacy assessments will also include changes in select co-morbidities, quality of life assessments, and changes in hunger and satiety, among others. Safety assessments include subject and investigator reported adverse events, physician follow-up assessments, and blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Potential subject was sham participant in the Essential pivotal trial
3. Potential subject agrees to be compliant with study and has a documented history of compliance in pivotal study.
4. Subjects between the ages of 23-61 years.
5. If female, be either post-menopausal, surgically sterile or agree to practice birth control during year of study and have negative serum HCG at screening/baseline.
6. Have a Body Mass Index (BMI) of ≥30 and <35 with at least one non-severe co-morbid obesity related condition or a BMI ≥ 35 with or without a non-severe obesity related co-morbid condition, where a severe co-morbid condition is defined as severe if symptoms cause severe discomfort, performance of daily activities is compromised, and/or condition is not entirely controlled with prescription drug therapy (See Section 14)
7. Absence of current severe systemic disease (including, but not limited to: coronary artery disease, chronic obstructive pulmonary disease, congestive heart failure, cancer, and chronic renal disease)
8. Agrees not to undergo any additional weight loss interventional procedures or liposuction for 12 months following study enrollment.
9. Agrees not to utilize any prescription or over the counter weight loss medications OR those that can suppress appetite/induce weight loss for 12 months following study enrollment (including all stimulant medication).
10. Be willing to cooperate with post-operative dietary recommendations and assessment tests.
11. Residing within a reasonable distance from the Investigator's treating office (~50 miles) and able and willing to travel to the Investigator's office to complete all routine follow-up visits.

Exclusion Criteria:

1. History of (or intra-operative evidence of) prior bariatric, gastric or esophageal surgery.
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endolumenal instruments or procedure execution.
3. Severe gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with drug therapy.
4. Large hiatal hernia (>3 cm) by history or as determined by pre-enrollment endoscopy.
5. Pancreatic insufficiency/disease.
6. History of gastroparesis or symptoms that would be suggestive of gastroparesis.
7. Pregnancy or plans of pregnancy in the next 12 months.
8. Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 1 month of Visit 1. Intranasal/inhaled steroids are acceptable.
9. History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis
10. History or present use of insulin or insulin derivatives for treatment of diabetes
11. Type II Diabetes Mellitus (as defined by HgbA1c >6.5%) for greater than 11 years at the time of enrollment
12. If smoker, plans to quit smoking in the year after enrollment
13. Portal hypertension and/or varices.
14. Significant abnormality identified during Visit 2 (enrollment visit) with endoscopy revealing large hiatal hernia, gastric/duodenal ulcer, gastric erosions, gastric outlet obstruction or stenosis, etc.
15. Patient has a history of drug or alcohol abuse or positive at screening for drugs of abuse.
16. Present or past history of psychosis, bipolar disease, or obsessive compulsive disorder after pre-enrollment history and medical /psychological assessment
17. Non-ambulatory or has significant impairment of mobility.
18. Known hormonal or genetic cause for obesity including untreated hypothyroidism (TSH >5.0 U/ml).
19. Participating in another clinical study except for Essential Study.
20. Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.

Ages: 23 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lavin, MD, Principal Investigator — Crescent City Surgical Centre
Locations (11):
- United States (11):
  - Shea Campus -Scottsdale Healthcare, Scottsdale, Arizona
  - University of Miami Hospital, Miami, Florida
  - Hamilton Medical Center, Dalton, Georgia
  - Northshore/Evanston Hospital, Evanston, Illinois
  - Crescent City Surgical, Metairie, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Fairview UMMC-University, Minneapolis, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - WA University School of Medicine, St Louis, Missouri
  - Lexington Medical Center, West Columbia, South Carolina
  - Baptist Memorial Hospital, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Essential Study Sham Cross-over: Eligible sham subjects from primary study
Period: Overall Study
Arm/Group | Essential Study Sham Cross-over
Started | 73
Completed | 50
Not Completed | 23
Not completed — Lost to Follow-up | 23

BASELINE CHARACTERISTICS:
Arm/Group | Essential Study Sham Cross-over
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Total Body Weight Loss
Description: Percent total body weight loss calculated through 12 months post procedure
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: percentage of TBW
Groups:
- Essential Study Sham Cross-over: This is a multicenter, un-blinded, open label, pivotal supplemental study to G130163 intended to evaluate the safety and efficacy of treating previous sham subjects in the Essential pivotal trial (IDE#G130163) with the active treatment (the placement of g-Cath EZ suture anchors along with diet and exercise). Compliant sham subjects (those who attended all primary IDE follow-up visits AND who continue to meet eligibility criteria as described in this protocol) will be offered this active treatment after their 12 month unblinding visit in the Essential pivotal trial.
Arm/Group | Essential Study Sham Cross-over
Number analyzed (Participants) | 50
percentage of TBW | 5.7 (6)

ADVERSE EVENTS:
Arm/Group | Essential Study Sham Cross-over
All-Cause Mortality (participants affected / at risk) | 0/73
Serious Adverse Events (participants affected / at risk) | 3/73
Other Adverse Events (participants affected / at risk) | 2/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essential Study Sham Cross-over (N=73)
Dehydration (General disorders) | 2 (2) — Procedure related event
Nausea (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Essential Study Sham Cross-over (N=73)
Kidney Infection (Renal and urinary disorders) | 2 (2) — Not related to device or procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No